CLINICAL TRIAL: NCT02487290
Title: Feasibility Study of Treatment Type II Endoleaks With ACP-T5: a Novel Approach.
Brief Title: ANEUFIX for Endoleaks Type II
Acronym: ACP-T5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TripleMed B.V. (Industry)
Collaborators: Fakkel bvba (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: TripleMed 001
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: AAA; Endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Intervention Model Description: This is a feasibility study, where initially 5 patients are to be treated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Aneufix ACP-T5
  Interventions: Device: Aneufix ACP-T5

INTERVENTIONS:
Device: Aneufix ACP-T5 — The ACP-T5 is injected via translumbar approach into the aneurysm sac near the entrance/exit of bloodvessel. ACP-T5 will cure and block the endoleak.
  Other Names: ANEUFIX

SUMMARY:
The study is a non-randomized, multi-center safety and feasibility trial of Aneufix ACP-T5 to treat patients with Isolated type II endoleak in the presence of a non-shrinking AAA sac following an EVAR procedure.

DETAILED DESCRIPTION:
The investigational device is called Aneufix, more specifically the model ACP-T5, which is a product treating the endoleak by blockage of backflowing blood vessels, i.e. by filling the 'endoleak void and nidus of feeding artery and exit of existing draining arteries'.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent type IIa or IIb endoleak (more than 6 months post-EVAR or post-embolization procedure); AND
2. Volume of the 'endoleak void' can be determined upfront; AND
3. An EVAR without circulatory complications; AND
4. An endoleak confirmed by CT scan in preceding 6 weeks demonstrating the high likelihood of the isolated nature of the endoleak; AND
5. An aneurysm sac growing in contours after EVAR (per European Guidelines) as documented in the preceding 6 weeks by means of echo (or alternative visualization technique); AND
6. An aneurysm sac that can be punctured in translumbar approach ; AND
7. Possibility to withhold anti-thrombogenic medication temporarily; AND
8. Ability and willingness to undergo the translumbar procedure under local anesthesia in a CT scan; AND
9. Be older than 18 years.

Exclusion Criteria:

1. Patient not able or willing to give written Informed Consent; OR
2. Patient undergoing emergency procedures; OR
3. Patient with traumatic vascular injury; OR
4. Patient with hemostatic disorder or who is clinically unstable; OR
5. Patient with a too high risk of abdominal sac rupture to allow safe radiological and scanographic assessments; OR
6. Patient who is allergic to contrast media or anticoagulants; OR
7. Patient with renal impairment (serum creatinine > 2 mg/dl or > 176 mmol/l); OR
8. Patient who is participating in another trial with an investigational drug or medical device; OR
9. Women of child-bearing potential; OR
10. Patient with a life expectancy of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Technical success of Type II endoleak repair with Aneufix ACP-T5 as demonstrated by the absence of an endoleak at the end of the procedure. | 24h
  At the end of the injection procedure, the technical success will be determined by angiographic recording and physician assessment of absence of endoleak. CT scan at 24 hrs is obtained to reconfirm the absence of endoleak.

SECONDARY OUTCOMES:
Clinical succes rate. | 6 and 12 months
  The clinical succes rate is defined as the absence of aneurysm sac growth after the procedure of ACP-T5 injection.
Safety aspects I : intra-operative complication rate. | All complications observed during the ACP-T5 injection procedure are documented.
  Intra-operative occurrence of complications.
Safety aspects II: Peri-operative complication rate. | 1 month
  All complications as well as the occurrence of adverse events and adverse device effects during the period of 24 hrs - 1 month are observed, documented, adjudicated and reported. adverse device effects are observed, documented, adjudicated and reported.
Safety aspects III : Mid- and long-term complication rate. | 1-12 months
  All complications as well as the occurrence of adverse events and adverse device effects during the period of 1-12 months are observed, documented, adjudicated and reported. adverse device effects are observed, documented, adjudicated and reported.
Aneurysm sac rupture. | 12 months
  The aneurysm sac rupture rate is assessed over a period of 12 months.
Survival. | 24 months.
  The survival rate throughout the study and up to 24 months is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eefting, Dr, Principal Investigator — Medisch Centrum Westeinde Den Haag; Erik Vermeulen, Dr, Principal Investigator — Spaarne Gasthuis, Haarlem
Locations (2):
- Netherlands (2):
  - Spaarne Gasthuisberg, Haarlem
  - Medisch Centrum Westeinde, The Hague

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share with other investigators then those participating in the study.

REFERENCES:
- [Derived] Smorenburg SPM, Lely RJ, Kelckhoven BV, Vermeulen EG, Yeung KK, Kruse RR, Kraai M, Stassen CM, Jacobs MJ, Hoksbergen AWJ. Initial Clinical Experience With AneuFix Injectable Biocompatible Elastomer for Translumbar Embolization of Type 2 Endoleaks. J Endovasc Ther. 2025 Feb;32(1):57-67. doi: 10.1177/15266028231165731. Epub 2023 Apr 19. PMID 37073926